CLINICAL TRIAL: NCT01109654
Title: A Prospective, Observational Study on the Use of Cetrotide (GnRH Antagonist) With GONAL-f in Assisted Reproductive Technologies (ART)
Brief Title: An Observational Study of Cetrotide® Gonadotropin-releasing Hormone Antagonist (GnRH Antagonist) With GONAL-f® in Assisted Reproductive Technologies (ART)
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Pte. Ltd., Singapore (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR200088-500
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2012-01

CONDITIONS: Infertility
Keywords: Fertilization in Vitro; Reproductive Techniques, Assisted; Follicle Stimulating Hormone; Cetrotide; Gonal-f
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — cetrorelix; follitropin alfa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, Serum, Tissue, Urine
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetrorelix acetate and Follitropin alfa — Cetrorelix acetate given either as a single-dose regimen of 3 mg injection or as a multiple-dose regimen of 0.25 mg daily injection.Ovarian stimulation therapy with Follitropin alfa generally starts on cycle Day 2 or 3. The starting dose of Follitropin alfa is based on the Investigators' discretion
  Other Names: Cetrotide; Gonal-f

SUMMARY:
This is a multicentric, prospective, observational study on the use of Cetrotide to control the endogenous gonadotrophin levels in Gonal-f stimulated ART treatment cycles in the Asia-Pacific region. The study plans to enrol approximately 1800-2000 subjects over a 9-month period at each participating centre.

This observational study is initiated to collect information on the use of Cetrotide (GnRH antagonist) in ART cycles in routine practice across the Asia-Pacific region. The information will allow a better understanding of the current ovarian stimulation regimens that involve Cetrotide in the control of the endogenous gonadotrophin concentrations. The collection of live birth data, though a challenging task, as a secondary endpoint will allow the study to show valuable information on the final objective of ART. To minimize the potential variability due to the different ovarian stimulation agents, the study is to include cycles treated with Gonal-f (recombinant human FSH) since this agent is widely available in the region.

DETAILED DESCRIPTION:
Gonadotrophin-releasing hormone (GnRH) antagonists were introduced in the beginning of this decade for the use in ART. The potential advantages of GnRH antagonists over the GnRH agonists include the avoidance of an acute stimulation of endogenous gonadotrophins and a dramatic reduction in the length of analogue treatment.

Despite the plus points of GnRH antagonists in ART, there has been some concern over the lower pregnancy rate reported, which may be the cause of a lower acceptance of GnRH antagonists in ovarian stimulation for in vitro fertilization (IVF). Interestingly, a separate meta-analysis did not reach the same finding. The probability of live birth after ovarian stimulation for IVF was found not to be dependent on the type of analogue used for pituitary suppression Cetrotide, a GnRH antagonist from Merck Serono, is currently approved for the inhibition of premature luteinizing hormone (LH) surges in women undergoing controlled ovarian stimulation in majority of the regions. It is given either as a single-dose regimen of 3 mg injection or as a multiple-dose regimen of 0.25 mg daily injection. Both regimens have been shown to offer equivalent efficacy and safety outcomes.

OBJECTIVES:

Primary objective:

* To assess the effectiveness of Cetrotide regimens, when used with Gonal-f, in routine ART treatment cycles

Secondary objectives:

* To assess the effectiveness of Cetrotide regimens on other efficacy endpoints
* To survey the types of Cetrotide regimen used and their success rates
* To assess the safety of Cetrotide regimens
* To explore the association between subject characteristics and treatment outcomes

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are undergoing ovarian stimulation for IVF or ICSI therapy
* Decision by treating physician to prescribe Gonal-f for controlled ovarian stimulation prior to study enrolment
* Decision by treating physician to prescribe Cetrotide as the down-regulation agent prior to study enrolment

Exclusion Criteria:

* Subjects using GnRH agonist as the down-regulation agent
* Contraindicated use of Cetrotide based on local label
* Subjects who have participated in the study previously
* Subjects with hypersensitivity to cetrorelix acetate, extrinsic peptide hormones or mannitol
* Subjects with known hypersensitivity to GnRH or any other GnRH analogs
* Subjects with known or suspected pregnancy, and lactation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Female subjects undergoing controlled ovarian stimulation.
Sampling Method: Non-Probability Sample
Enrollment: 2175 (Actual)
Dates: Start 2008-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving a clinical pregnancy. | At post hCG days 35-42
  A transvaginal ultrasound scan will be performed on all subjects who become pregnant provided that no miscarriage has occurred.

SECONDARY OUTCOMES:
Proportion of subjects with cancelled cycles | 3 month
Proportion of women with OHSS or risk of OHSS | 3 month
Duration and dose of Cetrotide administered | 3 month
Assessment of baseline characteristics | 3 month
  Assessment of subjects age, weight, height, FSH and LH level prior to Gonal-f administration, concomitant treatment, infertility history and infertility treatment
Total dose of Gonal-f administered | 3 month
Duration of ovarian stimulation | 3 month
Number of oocytes retrieved | 3 month
Number of subjects with Adverse Events | 3 month
Pregnancy rate | 12 month
Live birth rate | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Pte. Ltd., Singapore
Locations (1):
- Singapore General Hospital Pte Ltd, Outram Road, Singapore, Singapore